CLINICAL TRIAL: NCT06746870
Title: A Phase II Clinical Study to Evaluate the Safety, Pharmacokinetic Profile, and Preliminary Efficacy of IMM2510 in Combination with Chemotherapy As First-line Treatment in Subjects with Non-small Cell Lung Cancer or Triple-negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMM2510-003
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: NSCLC; TNBC
Keywords: NSCLC; TNBC; IMM2510
MeSH Terms: interventions — Drug Therapy; Pemetrexed; Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1a (Experimental): NSQ-NSCLC
  Interventions: Drug: IMM2510; Drug: Chemotherapy (pemetrexed + cisplatin/carboplatin)
- Cohort 1b (Experimental): SQ-NSCLC
  Interventions: Drug: IMM2510; Drug: Chemotherapy (paclitaxel + cisplatin/carboplatin)
- Cohort 2 (Experimental): TNBC
  Interventions: Drug: IMM2510; Drug: Chemotherapy(Nab-paclitaxel)

INTERVENTIONS:
Drug: IMM2510 — Cohort1:
  Phase I #: 10 mg/kg or 20 mg/kg, Q3W, intravenous infusion Phase II &: 20 mg/kg, Q3W, intravenous infusion
  Cohort2:
  Phase I #: 10 mg/kg or 20 mg/kg, Q2W, intravenous infusion Phase II &: 20 mg/kg, Q2W, intravenous infusion
Drug: Chemotherapy (pemetrexed + cisplatin/carboplatin) — Non-squamous non-small cell lung cancer (NQ-NSCLC): Pemetrexed 500 mg/m2 in combination with carboplatin (AUC 5-6) or cisplatin (75 mg/m2), intravenous infusion, Q3W, for 4 cycles, followed by maintenance treatment with pemetrexed
  Arms: Cohort 1a
Drug: Chemotherapy (paclitaxel + cisplatin/carboplatin) — Squamous non-small cell lung cancer (SQ-NSCLC): Paclitaxel 175 mg/m2 + carboplatin (AUC 5-6) or cisplatin (75 mg/m2), intravenous infusion, Q3W, for 4 cycles.
  Arms: Cohort 1b
Drug: Chemotherapy(Nab-paclitaxel) — Nab-paclitaxel, 100 mg/m2, 4 weeks as a cycle, administered on D1, 8, and 15 of each cycle.
  Arms: Cohort 2

SUMMARY:
This is a single-arm, multicenter, open-label Phase II clinical study evaluating the efficacy and safety of IMM2510 in combination with chemotherapy as first-line treatment in patients with stage IV metastatic or recurrent NSCLC or unresectable locally advanced or metastatic TNBC.

The target population includes: Cohort 1: Patients with histologically or cytologically confirmed stage IV metastatic or recurrent NSCLC who are EGFR wild-type and negative for ALK or ROS1 fusion genes, and who have not received prior systemic treatment for NSCLC; Cohort 2: Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic TNBC who are negative for estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor-2 (HER-2), and who have not received prior systemic treatment for TNBC; This study is divided into two phases. Phase I is the safety run-in period, which will preliminarily explore the safety and PK profile of IMM2510 in combination with chemotherapy in patients with NSCLC or TNBC who have previously failed at least first-line systemic treatment, are intolerant to, or not suitable for first-line systemic treatment, to determine the dose for the combination treatment. Phase II is the expanded enrollment period, which will enroll NSCLC patients (Cohort 1; where Cohort 1a is for NSQ-NSCLC and Cohort 1b is for SQ-NSCLC), or TNBC patients (Cohort 2), according to the dose for the combination treatment determined in Phase I, to further explore the preliminary clinical efficacy, safety, and PK profile of IMM2510 in combination with chemotherapy as first-line treatment in patients with NSCLC or TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily sign the ICF for this study ;
2. Aged ≥ 18 years old;
3. Cohort 1: NSCLC; EGFR wild-type and negative for ALK or ROS1 fusion genes. Cohort 1a: Non-squamous NSCLC (NSQ-NSCLC); Cohort 1b: Squamous NSCLC (SQ-NSCLC); Cohort 2: Breast cancer, negative for ER, PR, and HER-2. Definition of negative for ER and PR: IHC ER < 1%, IHC PR < 1%. Definition of negative for HER-2: IHC HER-2 (-) or (1+); for HER-2 (2+), FISH testing must be performed and the result must be negative;
4. Cohort 1: Previous systemic treatment for advanced NSCLC has not been received. If neoadjuvant and/or adjuvant treatment was previously received, the time from the completion of neoadjuvant and/or adjuvant treatment to the occurrence of recurrence/metastasis must be ≥ 12 months; Patients enrolled in the safety run-in period have previously failed at least first-line systemic treatment, are intolerant to, or not suitable for first-line systemic treatment for NSCLC; Cohort 2: Previous systemic treatment for advanced TNBC has not been received. If neoadjuvant and/or adjuvant treatment included taxane-based anti-tumor treatment, the time from the completion of taxane-based neoadjuvant and/or adjuvant treatment to the occurrence of recurrence/metastasis must be ≥ 12 months; Patients enrolled in the safety run-in period have previously failed at least first-line systemic treatment, are intolerant to, or not suitable for first-line systemic treatment for TNBC;
5. ECOG score of 0 or 1;
6. Have measurable lesions (according to RECIST 1.1).
7. Expected survival ≥ 12 weeks;
8. Provide archival tumor tissue samples or newly obtained needle biopsy or surgical resection samples of tumor lesions (previously unirradiated) for central PD-L1 and other biomarker tests. Formalin-fixed, paraffin-embedded (FFPE) tissue blocks are preferred over slides. Newly obtained biopsy samples are preferred over archival samples. Formalin-fixed samples are preferred after the subject is diagnosed with metastatic disease. If a recent biopsy is not feasible, biopsy samples obtained prior to adjuvant/neoadjuvant chemotherapy are acceptable.
9. Upon signing the ICF, females of childbearing potential and males must agree to practice effective contraception during the study and for 6 months after the last dose, and females of childbearing potential must have a negative result for pregnancy test within 3 days pre-dose;

Exclusion Criteria:

1. Received approved or investigational anti-tumor treatments within 4 weeks prior to the start of study treatment
2. Received nonspecific immunomodulatory treatments within 2 weeks prior to the start of study treatment;
3. Previously received any antibody or inhibitor targeting PD-1/PD-L1 or VEGF;
4. Laboratory abnormalities
5. History of pulmonary fibrosis or current presence of severe pulmonary functional impairment
6. Uncontrolled chronic disease
7. Unresolved toxicity
8. Uncontrolled brain metastases
9. Active infection
10. Bleeding Risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the preliminary clinical efficacy of IMM2510 for Injection in combination with chemotherapy as first-line treatment in patients with stage IV metastatic or recurrent non-small cell lung cancer (NSCLC) | 96 weeks
  Objective response rate for NSQ-NSCLC (ORR, assessed by the investigator) Objective response rate for SQ-NSCLC (ORR, assessed by the investigator)
To evaluate the preliminary clinical efficacy of IMM2510 for Injection in combination with nab-paclitaxel as first-line treatment in patients with unresectable locally advanced or metastatic triple-negative breast cancer (TNBC) | 96 weeks
  ORR (intention-to-treat (ITT), assessed by the investigator)

CONTACTS AND LOCATIONS:
Overall Officials: Qiying Lu, MD, Study Director — ImmuneOnco Biopharmaceuticals (Shanghai) Inc.

IPD SHARING:
Plan to Share IPD: No